CLINICAL TRIAL: NCT02408822
Title: Superiority of Drug-eluting Balloon Angioplasty Versus Plain Balloon Angioplasty for the Treatment of Hemodialysis Vascular Access Stenosis : a Multicentre, Randomized, Controlled Trial
Brief Title: Drug-Eluting Balloon Angioplasty for the Treatment of Hemodialysis Vascular Access Stenosis (DEBAVAS)
Acronym: B3AV
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-AOI-03
Record Dates: First submitted 2015-03-31; First posted 2015-04-06 (Estimated); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Dysfunction of Hemodialysis Vascular Access (Fistula and Graft)
MeSH Terms: conditions — Fistula

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PBA (Plain Balloon Angioplasty) (Active Comparator): Patient receiving endovascular treatment of a vascular access stenosis by plain balloon angioplasty (mechanical action, without drug)
  2-minutes inflation of the plain balloon on pre-dilated stenosis segment, at nominal pressure
  Interventions: Device: PTA Balloon dilatation catheter Advance® (Cook® Medical)
- PTX (Experimental): (PacliTaXel-coated balloon angioplasty) Patient receiving endovascular treatment of a vascular access stenosis by drug-eluting balloon angioplasty (mechanical action + antiproliferative drug - Paclitaxel) 2-minutes inflation of the drug-eluting balloon on pre-dilated stenosis segment, at nominal pressure
  Interventions: Device: Drug-eluting PTA Balloon dilatation catheter Advance® 18 PTX®

INTERVENTIONS:
Device: PTA Balloon dilatation catheter Advance® (Cook® Medical) — 2-minutes inflation of the plain balloon on pre-dilated stenosis segment, at nominal pressure
  Arms: PBA (Plain Balloon Angioplasty)
Device: Drug-eluting PTA Balloon dilatation catheter Advance® 18 PTX® — 2-minutes inflation of the drug-eluting balloon on pre-dilated stenosis segment, at nominal pressure
  Arms: PTX

SUMMARY:
Paclitaxel is an antiproliferative drug that can limit vascular intimal hyperplasia. Paclitaxel-coated balloons already have indications in the treatment of peripheral arterial disease.

This randomized controlled trial is designed to prove the superiority of a drug-eluting balloon catheter (Paclitaxel-coated balloon) over a plain balloon catheter in the treatment of stenosed autogeneous and prosthetic vascular accesses, in hemodialysis patients.

The hypothesis is that use of drug-eluting balloon will improve post-interventional patency of the access, and therefore, limit numbers and days of hospitalization for maintenance of hemodialysis vascular accesses.

DETAILED DESCRIPTION:
Introduction:

Half of patients with hemodialysis vascular access will present at least one episode of dysfunction within 1 year after creation, mainly due to intimal hyperplasia and stenosis. Paclitaxel is an antiproliferative drug that can limit intimal hyperplasia in vessels. Paclitaxel-coated balloons already have indications in the treatment of peripheral arterial disease.

Main objective:

To show that the use of Paclitaxel-coated balloons to treat stenosis of vascular accesses will improve post-interventional patency and reduce numbers and days of hospitalization for access maintenance in hemodialysis vascular access.

Hypothesis:

Paclitaxel-coated balloon angioplasty (PTX) prolongs primary patency of the access after treatment of vascular access stenosis compared to plain balloon angioplasty (PBA)(standard treatment).

Methodology:

We designed a prospective, single-blinded, multicenter, randomized, controlled trial, which aim to enroll 120 patients.

Patients diagnosed with a stenosis on their dysfunctional vascular access line (brachial-cephalic autogeneous fistula or brachial-axillary prosthetic graft) will be randomized to either arm of the study after completion of a successful pre-dilation with a standard plain balloon catheter.

Randomization will be stratified according to type of access (brachial-cephalic autogeneous fistula or brachial-axillary prosthetic graft).

Primary outcome measure will be primary patency of the vascular access at 12 months after treatment. Secondary outcome measures will be primary patency at 6 months, assisted-primary and secondary patencies at 6 and 12 months, number of re-interventions and number of days of hospitalization for re-intervention at 12 months.

Clinical significance:

By prolonging the vascular access lifespan, Paclitaxel-coated balloon angioplasty can limit morbidity and cost of vascular access maintenance for hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 years of age or older at the time of signing and dating informed consent (no upper age limit), can be male or female.
* Patient must have a vascular access for hemodialysis (type: brachial-cephalic autogeneous fistula or brachial-axillary prosthetic graft)
* Patient must have a dysfunction of its vascular access, defined by :

  * dialysis sessions last >4 hours
  * and/or access flow < 400ml/min for fistulae and <600ml for grafts, or 20% decrease in access flow as monitored during dialysis or by Duplex ultrasound scan,
  * and/or dialysis recirculation
  * and/or thrill not perceived
  * and/or pulsatile vascular access
  * and/or bleeding or increased bleeding time after puncture
* A stenosis >50% of the venous line must be diagnosed on the initial fistulogram
* A successful plain balloon angioplasty of the stenosis, defined by residual stenosis <30% on control angiogram, without dissection or indication for use of stent or additional surgical procedure, must be completed before inclusion.

Exclusion Criteria:

* Pregnant or nursing woman, or plans to become pregnant during the study.
* Patient has hyperkalemia >6,5 mmol/L with EKG modifications or acute cardiac insufficiency at the time of inclusion
* Vascular access has in-stent restenosis
* Initial fistulogram shows no stenosis
* Initial fistulogram shows indication for open surgical intervention
* Control fistulogram (after plain balloon angioplasty) shows indication for stenting or open surgical intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-09-29 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Primary patency of the vascular access after endovascular angioplasty of a stenosis with drug-eluting balloon compared with treatment with plain-balloon | at 12 months

SECONDARY OUTCOMES:
Primary patency of the vascular access | at 6 months after treatment
Assisted-primary patency of the vascular access | at 6 and 12 months after treatment
Secondary patency of the vascular access | at 6 and 12 months after treatment
Number of reinterventions (endovascular or surgery) | after treatment during the follow-up (at 12 months)
Days of hospitalization for reinterventions (endovascular or surgery) | after treatment during the follow-up (at 12 months)

CONTACTS AND LOCATIONS:
Overall Officials: REDA HASSEN-KHODJA, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (3):
- France (3):
  - CHU de Nice - Service de chirurgie vasculaire, Nice
  - Clinique St Georges, Nice
  - CHU de Reims, Reims